CLINICAL TRIAL: NCT05804448
Title: Effect of Altitude on Postdural Puncture Headache After Caesarean Delivery: a Prospective, Multicentre Cohort Study
Brief Title: Effect of Altitude on Postdural Puncture Headache After Caesarean Delivery
Status: Recruiting | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: Karnali Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Principal Investigator, B.P. Koirala Institute of Health Sciences
Other Study IDs: 533/2022 P
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Post-Dural Puncture Headache
Keywords: Spinal Anesthesia, Cesarean Section
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High-altitude group: Parturient who are native to their resident altitude, i.e. residing at the altitude above 2500 m from sea level will receive spinal anesthesia for caesarean section.
- Low-altitude group: Parturient who are native to their resident altitude, i.e. residing at the altitude below 500 m from sea level will receive spinal anesthesia for caesarean section.

SUMMARY:
The aim of this study is to examine the effects of altitude (high altitude versus low altitude) on incidence and severity of postural puncture headache (PDPH) following spinal anaesthesia for caesarean delivery. The investigators hypothesized that the risk of PDPH would be higher in highlander parturients than in lowlander parturients.

DETAILED DESCRIPTION:
This will be a prospective cohort study conducted in two different altitudes in Nepal. The high-altitude site is in Jumla, approximately 2514 m above the sea level, and a low altitude city is Dharan, located at 350 m from sea level.

The investigators will screen the eligible participant admitted to the in-patient obstetric unit. The investigator will also record patient baseline characteristics, preoperative anxiety, antenatal depression, presence of chronic pain conditions or preexisting headache. Spinal anaesthesia will be administered in the sitting position at the L3-L4 or L4-L5 interspace using a 25-G pencil point spinal needle (Pencan® 25-gauge).

The diagnosis of post-dural puncture headache will be based on the international headache society ICDH-3 criteria

ELIGIBILITY:
Inclusion Criteria:

* Parturient, aged more than or equal to 18 years
* American society of Anesthesiologist 2 and 3
* Scheduled for elective and non-elective (category 2 & 3) caesarean delivery with spinal anesthesia
* Native to their resident altitude i.e., those born, raised, and have continuously lived at the same altitude, at least for the past 1 year.

Exclusion Criteria:

* Hypertensive disorder
* Cerebrovascular disease
* Mental disorder (schizophrenia and other psychotic disorders)
* Known fetal anomalies
* Contraindication to spinal anaesthesia.
* Those requiring general anaesthesia for delivery due to failed spinal anesthesia
* Major post-delivery complications (severe haemorrhage, sepsis, or ICU admission)
* Those who migrate from their resident altitude (either low to high or vice versa) within 7 days post-delivery will also be excluded.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Parturients planned for elective and non-elective (category 2 & 3) caesarean section under spinal anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postdural puncture headache | up to 7 days after spinal anesthesia
  The diagnosis of post-dural puncture headache will be based on the international headache society ICDH-3 criteria: a headache that occurs within 5 days of a dural puncture, is located in the occipital and/or frontal areas, worsens within 15 min of sitting or standing and alleviates within 15 min after lying down, associated with at least one of the following features: neck stiffness, nausea, vomiting, photophobia, and tinnitus, and resolves either spontaneously within 1 week or within 48 h after effective treatment.

SECONDARY OUTCOMES:
Number of patients with severity of postdural puncture headache | up to 7 days after spinal anesthesia
  using a numeric rating scale (NRS), with 0= NO pain 10=worst imaginable pain, and classified as none (NRS=0), mild (1-3), moderate (4-6), and severe (7-10)
Number of patients with non-postdural puncture headache | up to 7 days after spinal anesthesia
  Headache that is not related to posture
Number of patients who received treatment for postdural puncture headache | up to 1 month after occurrence of PDPH
  paracetamol, NSAID's, caffeine, opioids, glossopharyngeal nerve block, sphenopalatine ganglion block and epidural blood patch

CONTACTS AND LOCATIONS:
Locations (2):
- Nepal (2):
  - Karnali Academy of Health Sciences, Jumla, Karnali
  - BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi